CLINICAL TRIAL: NCT00310999
Title: Comparison of Shikani Optical Scope to Macintosh Laryngoscope for Intubation of Patients With Potential Cervical Spine Injury
Brief Title: C-Spine Movement - Shikani Optical Scope vs Macintosh Laryngoscope for Patients With Cervical Spine Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R-05-400; REB #: 11688; CRIC R-05-400
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Wounds and Injuries
Keywords: Cervical Vertebrae; Intubation, Intratracheal; Laryngoscopes; Fluoroscopy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Shikani Optical Stylet

SUMMARY:
Patients undergoing surgery will have laryngoscopy performed using two widely accepted techniques - Macintosh Laryngoscope and Shikani Optical Scope. The techniques will be timed and compared for cervical spine movement using fluoroscopy.

DETAILED DESCRIPTION:
Approval for the study has been obtained from the Review Board for Health and Sciences Research Involving Human Subjects of the University of Western Ontario. Informed and written consent will be obtained from patients who are undergoing elective surgery requiring general anesthesia with endotracheal intubation. Preoperative clinical assessment of the patients will include routine airway evaluation of dentition, mouth opening, tongue size, Mallampati score, and neck mobility.

While awake, the patients will be placed on the operating room table with a rigid board under their head, neck, and torso in order to simulate the table on which patients involved in trauma are placed in the emergency room. In-line stabilization (ILS), as recommended by the ATLS guidelines, will be applied to maintain the patient's head in the neutral position and reduce neck movement during laryngoscopy.

After standard pre-oxygenation, anesthesia will be induced in routine fashion with 2-3 mg/kg propofol and 2-5 mcg/kg fentanyl; rocuronium 0.8 mg/kg will be administered to effect muscle paralysis. The patient will be then be ventilated with sevoflurane in 100% Oxygen via bag and mask for 3 minutes.

After the patient is anesthetized, a sealed envelope containing computer a generated random assignment will be opened. Laryngoscopy will then be performed two times, with the Macintosh laryngoscope and with the Shikani Optical Scope, in random order as determined by the envelope. Between laryngoscopies, the patient will be ventilated with sevoflurane in 100% Oxygen.

For direct Macintosh laryngoscopy, a size 3 laryngoscope blade will be recommended in all patients. With laryngoscopy, the glottis will be exposed to enable positioning of the endotracheal tube at the vocal cords. During the second laryngoscopy in the above sequence, the trachea will be intubated.

The study is then complete. The hard board will be removed and the surgery will proceed in the usual fashion.

The laryngoscopy and intubation will be recorded by a portable fluoroscopy unit for subsequent review by the radiologist to assess relative neck movement.

Laryngoscopy time will be defined as the time from when the laryngoscope blade or Shikani stylet passes the teeth of the patient until the time the endotracheal tube is positioned at the opening of the larynx. If the intubation sequence is longer than 120 seconds, it will be deemed a failure and recorded as such.

The Cormack (11) of the larynx will be recorded for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective non-cardiac surgery patients requiring intubation for the surgery.
* Age 18-75
* ASA 1-3
* Body Mass Index (BMI) < 40

Exclusion Criteria:

* patients with previous neck surgery or unstable C-spine
* patients with Reflux disease (GERD)
* patients who are or may be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-03 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
cervical spine movement

SECONDARY OUTCOMES:
Duration of intubation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, MD, Principal Investigator — London Health Sciences Centre; Rosemary A Craen, MD, Principal Investigator — London Health Sciences Centre; David M Pelz, MD, Principal Investigator — London Health Sciences Centre; Allison Shakih, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre University Hospital Site, London, Ontario, Canada

REFERENCES:
- [Background] Turkstra TP, Craen RA, Pelz DM, Gelb AW. Cervical spine motion: a fluoroscopic comparison during intubation with lighted stylet, GlideScope, and Macintosh laryngoscope. Anesth Analg. 2005 Sep;101(3):910-915. doi: 10.1213/01.ane.0000166975.38649.27. PMID 16116013
- [Background] Sawin PD, Todd MM, Traynelis VC, Farrell SB, Nader A, Sato Y, Clausen JD, Goel VK. Cervical spine motion with direct laryngoscopy and orotracheal intubation. An in vivo cinefluoroscopic study of subjects without cervical abnormality. Anesthesiology. 1996 Jul;85(1):26-36. doi: 10.1097/00000542-199607000-00005. PMID 8694378
- [Background] Watts AD, Gelb AW, Bach DB, Pelz DM. Comparison of the Bullard and Macintosh laryngoscopes for endotracheal intubation of patients with a potential cervical spine injury. Anesthesiology. 1997 Dec;87(6):1335-42. doi: 10.1097/00000542-199712000-00012. PMID 9416718